CLINICAL TRIAL: NCT04236284
Title: Management of Chronic Pain and PTSD in Gulf War Veterans With tDCS+Prolonged Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Melba Hernandez-Tejada, PhD, DHA, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-19-0960
Record Dates: First submitted 2020-01-14; First posted 2020-01-22 (Actual); Results first posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Chronic Pain; PTSD
MeSH Terms: conditions — Chronic Pain; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Home-based tDCS + Prolonged Exposure Therapy (Experimental): Participants will come in person to the clinic office to complete the baseline visit and the in-person training for the use of both home-based self-administered tDCS and the home-based telehealth device (iPad) for the PE sessions. They understand that they will start the sessions of tDCS once they start the in vivo and imaginal exposures assignments at home. They will self-administer (under televideo supervision) the tDCS session before doing in vivo and/or imaginal exposures assignments. The participants will be remotely supervised by trained research staff at each stimulation to ensure the technique is correct and to monitor any adverse events. We will provide secure videoconferencing software (e.g., WebEx) and ensure the participants are comfortable using the telehealth software.
  Interventions: Device: Home-based tDCS; Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Device: Home-based tDCS — tDCS is a non-invasive neuromodulation technique that has been used to improved cognitive functions. It will be administered with a constant current intensity of 2 mA57 for 20 min per session/ 10 sessions total daily for 2 weeks (Monday to Friday). The device is a Soterix 1x1 tDCS mini-CT Stimulator (Soterix Medical Inc., NY) with headgear and 5 _ 7 cm saline-soaked surface sponge electrodes.
  Other Names: Soterix 1x1 tDCS mini-CT Stimulator
Behavioral: Prolonged Exposure Therapy — Prolonged Exposure Therapy is a treatment for PTSD that includes the following components: a) psycho-education about the common reactions to traumatic events and presentation of the treatment rationale (sessions 1 and 2), b) repeated in vivo exposure to traumatic stimuli (in vivo exercises are assigned as homework during sessions 3 through 11), c) repeated, prolonged, imaginal exposure to traumatic memories (imaginal exposure is implemented during sessions 3 through 11; patients listen to session audiotapes for homework between sessions), and d) relapse prevention strategies and further treatment planning (session 12).

SUMMARY:
Gulf War Veterans (a DoD/VA defined service era corresponding to the first Gulf War under operations Desert Storm and Desert Shield 1990-1991), especially those who present with Post-Traumatic Stress Disorder (PTSD), are particularly likely to experience chronic pain. Veterans with co-morbid chronic pain and PTSD utilize healthcare services at a higher rate than those with pain or PTSD alone. Unfortunately, there are no integrated treatments for Pain and PTSD. Moreover, non-pharmacological treatments for pain such as Cognitive Behavioral Therapy are useful in only about 50% of cases. Transcranial direct current stimulation (tDCS) may be an effective treatment for pain, and has been recently used to ameliorate PTSD symptoms. Prolonged Exposure Therapy (PE) is highly effective in treating PTSD symptoms. Therefore, we propose to (a) integrate & (b) gather feasibility data for home-based tDCS + PE for Pain and PTSD with 15 Gulf War Veterans.

The Overall Aim of the present proposal is to integrate, refine and investigate the feasibility (e.g., pilot testing, recruitment, attrition, assessment) of tDCS for treating chronic pain with a best practices evidence-based treatment for PTSD (i.e., Prolonged Exposure: PE) in 15 Gulf War veterans, a group for which both pain (fibromyalgia) and PTSD are particularly problematic.

DETAILED DESCRIPTION:
Chronic pain is one of the most prevalent health conditions among Americans, affecting about a third of the general population. In Gulf War (1990-1991) veterans, chronic pain is even more common, with a prevalence of about 50%. Indeed, the pain-related fibromyalgia diagnosis is part of Gulf War Syndrome and is highly comorbid with other common military service-related health problems such as Posttraumatic Stress Disorder (PTSD). Moreover, lack of effective, integrated, and available alternative treatments for chronic pain contributes to the opioid epidemic.

PTSD is also highly prevalent in Gulf War Veterans, at about 15-25% of Operation Desert Shield and Desert Storm Veterans. Moreover, several investigators note that PTSD treatment response is poorer for Veterans who experience chronic pain and for Veterans who served in the Gulf War.

The Overall Aim of the present proposal is to integrate, refine and investigate the feasibility (e.g., pilot testing, recruitment, attrition, assessment) of tDCS for treating chronic pain with a best practices evidence-based treatment for PTSD (i.e., Prolonged Exposure: PE) in 15 Gulf War veterans, a group for which both pain (fibromyalgia) and PTSD are particularly problematic.

SA1: Integrate the home-based tDCS+PE Treatment. The investigative team is comprised of Pain, PTSD, and salivary biomarker experts who will integrate tDCS into the 12 session PE treatment protocol.

H1: The 12 session PE protocol will yield itself well to tDCS component integration based on participant feedback.

SA2: Test the feasibility of both the integrated intervention and key study design features, including translational research features such as biomarker assessment in a non-randomized trial with 15 Gulf War Veterans assessed at baseline and post-treatment. Feasibility of the home-based tDCS+PE intervention will be measured in terms of recruitment metrics, assessment burden, successful biomarker collection, specification of biomarker relationship to hypothesized mechanisms of change, treatment attrition, rates of missing data at each measurement time point, participant satisfaction, and ratings of treatment face validity. Post treatment key informant interviews will be conducted where suggestions for treatment enhancement and satisfaction will be systematically collected and analyzed.

H2 is given in terms of Specific Pre-Defined Milestones for Success, including: 75% of Veterans experiencing chronic pain (fibromyalgia) and PTSD who enroll will complete at least 8 sessions of the integrated treatment, and both completers and dropouts will offer actionable suggestions in exit interviews for improving the delivery of the intervention. SA2) Feasibility metrics will be acceptable for recruitment rate (two per month), treatment completion of 8 sessions (75%), assessment completion (90%), and good to excellent satisfaction (95%)

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic non-cancer pain and pain interference, defined as scoring 1 standard deviation above PROMIS normative data on both the 3-item PROMIS Pain Intensity 3a scal and the 8-item PROMIS Pain 8a Interference scale. Symptoms will be required to be of six-month duration or longer
* Diagnosis of PTSD assigned on the basis of the Clinician Administered PTSD Scale.

Exclusion Criteria:

* Having a household member who is already enrolled in the study
* Active psychosis or dementia at screening
* Suicidal ideation with clear intent
* Current substance dependence
* current opioid medication for pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melba Hernandez Tejada, PhD, DHA, Principal Investigator — UTHealth at Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hernandez-Tejada MA, Cherry KE, Rauch SAM, Acierno R, Fries GR, Muzzy W, Teng EJ, Wangelin B, Ahn H. Management of Chronic Pain and PTSD in Veterans With tDCS+Prolonged Exposure: A Pilot Study. Mil Med. 2023 Nov 3;188(11-12):3316-3321. doi: 10.1093/milmed/usac200. PMID 35808998

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Started | 21
Completed tDCS | 16
Completed Prolonged Exposure Therapy | 14
Completed | 14
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 8
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment as Assessed by Number of Participants Enrolled in the Study
Time Frame: Week 0
Measure: Count of Participants; unit: Participants
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 21
Participants | 21

2. Primary Outcome: Feasibility of Biomarker Collection as Assessed by Number of Planned Saliva Samples Divided by Number of Planned Saliva Samples Collected
Time Frame: Week 12
Population: Data were not collected for this outcome measure due to COVID restrictions.
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 0

3. Primary Outcome: Feasibility of Biomarker Viability as Assessed by Percent of Viable Saliva Samples
Time Frame: Week 12
Population: Data were not collected for this outcome measure due to COVID restrictions.
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 0

4. Primary Outcome: Feasibility of Retention as Assessed by Number of Participants Who Complete at Least 8 Sessions
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
Participants | 16

5. Primary Outcome: Feasibility of Data Collection as Assessed by Percent of Missing Data
Time Frame: Week 12
Measure: Number; unit: percentage of missing data
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
percentage of missing data | 0

6. Primary Outcome: Feasibility as Indicated by Satisfaction as Assessed by the Charleston Psychiatric Outpatient Satisfaction Scale
Description: The Charleston Psychiatric Outpatient Satisfaction Scale total score ranges from 13 to 65, with a higher score indicating higher satisfaction.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 42.48 (4.75)

7. Primary Outcome: Feasibility as Indicated by Treatment Credibility as Assessed by a Credibility Scale
Description: Treatment credibility will be assessed by a scale, with a total score ranging from 0 to 10, with 0 being "not credible, I did not think this treatment would help either my PTSD or Pain symptoms" to 10 being "completely credible, I was very sure this treatment would help both my PTSD and Pain symptoms."
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 8.9 (0.85)

8. Primary Outcome: Feasibility as Indicated by Treatment Acceptability as Assessed by an Acceptability Scale
Description: Treatment acceptability will be assessed by a scale, with a total score ranging from 0 to 10, with 0 being "not acceptable, this treatment should not be offered to veterans, those in pain, or those with PTSD" to 10 being "completely acceptable, this treatment is perfectly suited to veterans and others with pain and PTSD symptoms."
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 8.9 (0.85)

9. Primary Outcome: Pain Interference as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain 8a Interference Scale
Description: PROMIS Pain interference 8a assesses self-reported consequences of pain on relevant aspects of one's life in the past 7 days. The measure includes 8-items rating pain from "Not at all" = 1 to "Very much" = 5, therefore the response range is 8-40 with higher scores indicating greater pain interference.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 31.81 (4.05)

10. Primary Outcome: Pain Interference as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain 8a Interference Scale
Description: as for outcome 9
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 28.94 (7.32)

11. Primary Outcome: Pain Interference as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain 8a Interference Scale
Description: as for outcome 9
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 25.75 (8.69)

12. Primary Outcome: Pain Intensity as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain 3a Intensity Scale
Description: PROMIS Pain intensity 3a is a self-report measure that assesses how much a person hurts (intensity or severity) in the past 7 days. The measure includes three items rating pain from "Had no pain" = 1 to "Very severe" = 5, therefore the response range is 3-15 with higher scores indicating greater pain intensity. Raw scores are reported.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 11.19 (1.76)

13. Primary Outcome: Pain Intensity as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain 3a Intensity Scale
Description: as for outcome 12
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 10.50 (1.86)

14. Primary Outcome: Pain Intensity as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain 3a Intensity Scale
Description: as for outcome 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 10.25 (2.29)

15. Primary Outcome: PTSD Intensity as Assessed by the Clinician-Administered PTSD Scale 5 (CAPS-5)
Description: Total possible scores on the CAPS-5 scale range from 0 to 80, with a higher score indicating greater PTSD intensity.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 38.88 (9.01)

16. Primary Outcome: PTSD Intensity as Assessed by the Clinician-Administered PTSD Scale 5 (CAPS-5)
Description: Total possible scores on the CAPS-5 scale range from 0 to 80, with a higher score indicating greater PTSD intensity.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 33.93 (11.52)

17. Primary Outcome: PTSD Intensity as Assessed by the Clinician-Administered PTSD Scale 5 (CAPS-5)
Description: Total possible scores on the CAPS-5 scale range from 0 to 80, with a higher score indicating greater PTSD intensity.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 28.19 (14.05)

18. Secondary Outcome: PTSD as Assessed by the PTSD Checklist-5 (PCL-5)
Description: PCL-5 score ranges from 0 to 80, with a higher score indicating greater PTSD.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 57.69 (12.67)

19. Secondary Outcome: PTSD as Assessed by the PTSD Checklist-5 (PCL-5)
Description: PCL-5 score ranges from 0 to 80, with a higher score indicating greater PTSD.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 51.23 (14.20)

20. Secondary Outcome: PTSD as Assessed by the PTSD Checklist-5 (PCL-5)
Description: PCL-5 score ranges from 0 to 80, with a higher score indicating greater PTSD.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 38.33 (20.61)

21. Secondary Outcome: Depression as Assessed by the Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 score ranges from 0 to 27, with a higher score indicating greater depression.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 17.75 (4.77)

22. Secondary Outcome: Depression as Assessed by the Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 score ranges from 0 to 27, with a higher score indicating greater depression.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 17.31 (4.96)

23. Secondary Outcome: Depression as Assessed by the Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 score ranges from 0 to 27, with a higher score indicating greater depression.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 13.47 (6.37)

24. Secondary Outcome: Quality of Life as Assessed by the World Health Organization Quality of Life - Short Form (WHOQOL-BREF)
Description: There are 4 domains on the WHOQOL-BREF, listed below, and for all domains a higher score indicates a greater quality of life.
  * physical health domain (7 items) - total score ranges from 7 to 35
  * psychological health domain (6 items) - total score ranges from 6 to 30
  * social relationships domain (3 items) 3 - total score ranges from 3 to 15
  * environmental health domain (8 items) - total score ranges 8 to 40
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale
  physical health domain | 19.25 (2.67)
  psychological health domain | 15.33 (4.29)
  social relationships domain | 6.50 (2.91)
  environmental health domain | 25.18 (5.47)

25. Secondary Outcome: Quality of Life as Assessed by the World Health Organization Quality of Life - Short Form (WHOQOL-BREF)
Description: as for outcome 24
Time Frame: Week 6
Population: Data were not collected for this outcome measure.
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 0

26. Secondary Outcome: Quality of Life as Assessed by the World Health Organization Quality of Life - Short Form (WHOQOL-BREF)
Description: as for outcome 24
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale
  physical health domain | 20.50 (3.03)
  psychological health domain | 16.83 (3.16)
  social relationships domain | 8.00 (3.38)
  environmental health domain | 27.64 (5.45)

27. Secondary Outcome: Pain as Assessed by the West Haven-Yale Multidimensional Pain Inventory (WHYMPI/MPI)
Description: There are 13 subscales of the West Haven-Yale Multidimensional Pain Inventory (WHYMPI/MPI), with each subscale ranging in score from 0 to 6, with a higher score indicating a greater degree of the domain assessed by the subscale.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale
  Pain Interference | 4.73 (0.80)
  Support | 4.21 (1.70)
  Pain Severity | 4.54 (0.83)
  Perception of Control | 3.31 (1.16)
  Affective Distress | 4.21 (0.91)
  Negative Responses | 2.50 (1.34)
  Solicitous Responses | 2.42 (1.36)
  Distracting Responses | 2.38 (1.72)
  Household Chores | 3.10 (1.65)
  Outdoor Work | 2.03 (1.58)
  Activities away from Home | 2.00 (0.90)
  Social Activities | 2.13 (0.99)
  General Activity | 2.34 (0.93)

28. Secondary Outcome: Pain as Assessed by the West Haven-Yale Multidimensional Pain Inventory (WHYMPI/MPI)
Description: as for outcome 27
Time Frame: Week 6
Population: Data were not collected for this outcome measure.
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 0

29. Secondary Outcome: Pain as Assessed by the West Haven-Yale Multidimensional Pain Inventory (WHYMPI/MPI)
Description: as for outcome 27
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale
  Pain Interference | 4.09 (1.34)
  Support | 3.75 (1.35)
  Pain Severity | 3.75 (0.94)
  Perception of Control | 3.31 (1.46)
  Affective Distress | 3.50 (0.73)
  Negative Responses | 2.81 (1.27)
  Solicitous Responses | 3.17 (0.97)
  Distracting Responses | 3.25 (1.69)
  Household Chores | 2.68 (1.44)
  Outdoor Work | 2.53 (1.52)
  Activities away from Home | 2.47 (1.52)
  Social Activities | 2.47 (1.36)
  General Activity | 2.54 (1.30)

30. Secondary Outcome: Kinesiophobia as Assessed by the Tampa Scale of Kinesiophobia-Revised (TSK-R)
Description: Total score ranges from 17 - 68. A score of 17 is the lowest possible score, and indicates no kinesiophobia (that is, fear of pain with movement) or negligible kinesiophobia. A score of 68 is the highest possible score and indicates extreme kinesiophobia.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 46.64 (9.43)

31. Secondary Outcome: Kinesiophobia as Assessed by the Tampa Scale of Kinesiophobia-Revised (TSK-R)
Description: as for outcome 30
Time Frame: Week 6
Population: Data were not collected for this outcome measure.
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 0

32. Secondary Outcome: Kinesiophobia as Assessed by the Tampa Scale of Kinesiophobia-Revised (TSK-R)
Description: as for outcome 30
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 46.46 (11.78)

33. Secondary Outcome: Pain Catastrophizing as Assessed by the Pain Catastrophizing Scale (PCS)
Description: Total scores ranges from 0 to 52, with a higher score indicating greater Pain Catastrophizing.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 33.42 (11.27)

34. Secondary Outcome: Pain Catastrophizing as Assessed by the Pain Catastrophizing Scale (PCS)
Description: Total scores ranges from 0 to 52, with a higher score indicating greater Pain Catastrophizing.
Time Frame: Week 6
Population: Data were not collected for this outcome measure.
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 0

35. Secondary Outcome: Pain Catastrophizing as Assessed by the Pain Catastrophizing Scale (PCS)
Description: Total scores ranges from 0 to 52, with a higher score indicating greater Pain Catastrophizing.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 16
score on a scale | 29.42 (15.03)

36. Secondary Outcome: Salivary Biomarker Measurement
Description: Salivary levels of the biomarker panel (cortisol, substance P, DHEA, IL-1, and IL-6) using enzyme-linked immunosorbent assays (ELISA).
Time Frame: Week 0
Population: Data were not collected for this outcome measure due to COVID restrictions.
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 0

37. Secondary Outcome: Salivary Biomarker Measurement
Description: as for outcome 36
Time Frame: Week 6
Population: Data were not collected for this outcome measure due to COVID restrictions.
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 0

38. Secondary Outcome: Salivary Biomarker Measurement
Description: as for outcome 36
Time Frame: Week 12
Population: Data were not collected for this outcome measure due to COVID restrictions.
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Home-based tDCS + Prolonged Exposure Therapy
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT04236284/Prot_SAP_001.pdf